CLINICAL TRIAL: NCT05997160
Title: Research on Vaginal Microbiota Evaluation Unified Standards Based on Gram Staining
Acronym: VENUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Jiangsu Bioperfectus Technologies Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Fengxia Xue, Director of the Medical Center for Obstetrics and Gynecology, Tianjin Medical University General Hospital
Other Study IDs: IRB2023-YX-022-01
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospital name + infection type + number: There is no intervention.

SUMMARY:
The goal of this observational study is to explore a standardized sample process for improving the accuracy of vaginal microbiota evaluation and to explore a more complete and comprehensive method for vaginal microbiota evaluation based on gram staining.

DETAILED DESCRIPTION:
This study consists of two sub-studies:

1. Sub-study on Standardized method of Microscopic Slide Preparation: this sub-study aims to compare different slide preparation methods and dilution levels based on various aspects, including uniformity, impurities, clarity and so on, and then explore the optimal method and dilution level. Additionally, it will summarize the conversion method for white blood cells between wet mount and gram staining, and for white blood cells between high-power microscopy and oil immersion microscopy.
2. Sub-study on Vaginal Microbiota Evaluation on Gram Staining: For patients with diagnosed vaginal infection type, it will calculate the consistency of results between different laboratories. And it will evaluate the effectiveness combined artificial intelligence technology and other technological platforms. Besides, for patients without diagnosed vaginal infection type, different methods such as 16S rRNA gene sequencing and metagenomic sequencing are used for analysis and profiling to guide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women who visit our research settings and conduct vaginal discharge examination based on Gram-stained smear.
* No sexual intercourse, vaginal douching, or vaginal medication within the last 72 hours.
* Not during menstruation (menstrual period ended ≥3 days ago).

exclusion Criteria:

* Receiving systemic or vaginal antifungal or antibiotic treatment within the past week.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: VENUS study plans to enrol 5590 participants, aged 15-49 years, from visiting our research settings across the country who evaluate vaginal discharge based on Gram-stained smear.
Sampling Method: Non-Probability Sample
Enrollment: 5590 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The score for smear | December 2023
  This score consists of uniformity, impurities, cell degeneration, and clarity for evaluating a smear.
Diagnosis of vaginitis type | March 2024
  The Diagnosis of vaginitis type based on Gram-stained smear and antigen testing, including aerobic vaginitis(AV), bacterial vaginosis (BV), vulvovaginal candidiasis (VVC), trichomonal vaginitis (TV), and normal.
Relative Abundance | May 2024
  Relative Abundance is from 16S rRNA gene sequencing and metagenomic sequencing for patients without clearly diagnosis.
Intensity | May 2024
  The intensity is tested by liquid chromatography-tandem mass spectrometry for targeted metabolites for patients without clearly diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Fengxia Xue, PhD, Principal Investigator — Tianjin Medical University General Hospital